CLINICAL TRIAL: NCT05449782
Title: Proof-of-concept Study to Investigate Hand and Foot Microvascular Response to Cocoa Flavanols in Healthy and Type 2 Diabetes Participant
Brief Title: Macro- and Microvascular Response to Cocoa Flavanols in Healthy and Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: OCTA2
Record Dates: First submitted 2021-05-18; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-05

CONDITIONS: Microangiopathy, Diabetic; Polyphenol; Optical Tomography; Vascular Endothelium; Arterial Stiffness; Healthy Participants
MeSH Terms: conditions — Diabetic Angiopathies

STUDY DESIGN:
Intervention Model Description: 2 group (healthy and type 2 diabetes) randomised controlled cross-over (2-period, 2-sequence) study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Placebo and cocoa flavanols will be delivered in same number of identical appearing capsules
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy participants: Cocoa flavanol - Placebo (Other): Healthy participants receiving cocoa flavanols on first study day and placebo on second study day
  Interventions: Dietary Supplement: Cocoa flavanol; Other: Placebo
- Healthy participant: Placebo - Cocoa flavanol (Other): Healthy participants receiving placebo on first study day and cocoa flavanols on second study day
  Interventions: Dietary Supplement: Cocoa flavanol; Other: Placebo
- Type 2 diabetes participants: Cocoa flavanol - Placebo (Other): Participants with type 2 diabetes receiving cocoa flavanols on first study day and placebo on second study day
  Interventions: Dietary Supplement: Cocoa flavanol; Other: Placebo
- Type 2 diabetes participants: Placebo - Cocoa flavanol (Other): Participants with type 2 diabetes receiving placebo on first study day and cocoa flavanols on second study day
  Interventions: Dietary Supplement: Cocoa flavanol; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Cocoa flavanol — Commercially available Cocoa Via Brand capsules containing 1350 mg cocoa flavanols (6 capsules)
Other: Placebo — Capsules identical to ccocoa flavanol capsules filled with calorically matched brown sugar (6 capsules)

SUMMARY:
The greatest challenge in our ageing society are cardiovascular diseases such as stroke, heart attack, peripheral artery disease of the legs with non-healing wounds (ulcers), or diabetes. Specific diets with high polyphenol content are associated with lower incidence of cardiovascular disease and can improve macrovascular function when consumed acutely and chronically. Which role the smallest blood vessels (microcirculation) play in this and if the microcirculation responds to therapies is not well understood. One reason for this is that no generally available medical instrument has the resolution to study the microcirculation. The recently developed optical coherence tomography angiography (OCTA), currently mainly used by eye doctors, is able to visualise the microcirculation.

The current randomised controlled cross-over proof-of-concept study will test the acute effect of a cocoa flavanol intervention on cutaneous microvascular structure and function of hands and feet together with macrovascular function of upper and lower extremities in healthy and type 2 diabetes participants. It is the hypothesis that cocoa flavanol intervention as compared to placebo can acutely increase microvascular vasodilation and macrovascular endothelial function in arms and legs together with arterial stiffness in both healthy and type 2 diabetes participants.

ELIGIBILITY:
Healthy:

Inclusion Criteria:

* Healthy, 20-70 years
* BMI 20-30 kg/m^2

Exclusion Criteria:

* Diabetes mellitus
* Symptoms of acute infection
* Cardiac rhythm other than sinus
* Active malignancy
* Clinical signs or symptoms of cardiovascular disease (coronary artery disease, lower extremity artery disease, cerebrovascular disease): angina pectoris, dyspnea, palpitation, syncope, claudication
* Active vasoactive medication.

Type 2 Diabetes:

Inclusion Criteria:

* Type 2 diabetes mellitus
* 20-70 years
* BMI 20-30 kg/m^2

Exclusion Criteria:

* Symptoms of acute infection
* Cardiac rhythm other than sinus
* Active malignancy
* Clinical signs or symptoms of cardiovascular disease (coronary artery disease, lower extremity artery disease, cerebrovascular disease): angina pectoris, dyspnea, palpitation, syncope, claudication
* Active vasoactive medication.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Microvascular dilation | Change at 2 hours as compared to baseline after ingestion of cocoa flavanol vs placebo
  Microvascular diameter increase in response to 5 min limb occlusion on hands and feet
Macrovascular endothelial function | Change at 2 hours as compared to baseline after ingestion of cocoa flavanol vs placebo
  Flow-mediated dilation determined with ultrasound in brachial and common femoral artery

SECONDARY OUTCOMES:
Arterial stiffness | Change at 2 hours as compared to baseline after ingestion of cocoa flavanol vs placebo
  Pulse wave velocity (Arteriograph)
Blood pressure | Change at 2 hours as compared to baseline after ingestion of cocoa flavanol vs placebo
  Upper arm blood pressure measured with Arteriograph
Leg perfusion pressure | Change at 2 hours as compared to baseline after ingestion of cocoa flavanol vs placebo
  Doppler based perfusion pressure of leg

OTHER OUTCOMES:
Photoplethysmography (PPG) based pulse wave velocity (PWV) | Change at 2 hours as compared to baseline after ingestion of cocoa flavanol vs placebo
  PWV velocity calculated based on PPG sensor at hand and foot
Photoplethysmography (PPG) blood flow | Change at 2 hours as compared to baseline after ingestion of cocoa flavanol vs placebo
  Based on PPG signals on hand and foot

CONTACTS AND LOCATIONS:
Overall Officials: Christian Heiss, Prof., Principal Investigator — University of Surrey, Department of Clinical and Experimental Medicine
Locations (1):
- University of Surrey, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Will be decided on an individual basis and after study completion.